CLINICAL TRIAL: NCT01856712
Title: Pharmacotherapeutic Intervention to Improve Treatment Engagement Among Alcohol-dependent Veterans After Hospital Discharge
Brief Title: Oral vs. Injectable Naltrexone for Hospitalized Veterans With Alcohol Dependence
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0702
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Alcohol Dependence
Keywords: alcohol; veterans
MeSH Terms: conditions — Alcoholism | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral naltrexone (Active Comparator): an initial 50 mg oral dose of naltrexone prior to hospital discharge plus a 30-day prescription for oral naltrexone
  Interventions: Drug: Naltrexone
- injectable naltrexone (Experimental): a single 380 mg intramuscular injection of naltrexone (duration of action = 30 days)prior to hospital discharge followed by a second injection one month later.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Naltexone was chosen for this study because naltrexone is the only medication available in both oral daily and injectable monthly formulations, which will allow the study to examine issues around medication adherence.
  Other Names: Revia, Vivitrol

SUMMARY:
The over-arching goal of the proposed project is to understand the impact of medication adherence upon engagement in behavioral treatment for alcohol use disorders. The proposed project is a pilot feasibility study of inpatient veterans with problem alcohol use at the William S. Middleton VA Hospital (Madison, WI). Participants will be randomized to one of two parallel study conditions: (1) an initial 50 mg oral dose of naltrexone prior to hospital discharge plus a 30-day prescription for oral naltrexone, or (2) a single 380 mg intramuscular injection of naltrexone administered prior to discharge and a second injection one month later. The central hypothesis is that hospital-administered injectable naltrexone, when compared to daily oral naltrexone taken at home, will reduce alcohol use in the days immediately following hospitalization. Injectable naltrexone has been efficacious vs. placebo in addition to behavioral treatment in several studies. However, it has yet to be examined in head-to-head comparison with oral naltrexone, or in the hospital setting as an intervention that might facilitate behavioral treatment follow up after discharge.

DETAILED DESCRIPTION:
The proposed project is a pilot feasibility study of inpatient veterans with problem alcohol use at the William S. Middleton VA Hospital. The over-arching goal is to understand the impact of medication adherence upon engagement in behavioral treatment for alcohol use disorders. Participants will be randomized to one of two parallel study conditions: (1) an initial 50 mg oral dose of naltrexone prior to hospital discharge plus a 30-day prescription for oral naltrexone, or (2) a single 380 mg intramuscular injection of naltrexone (duration of action = 30 days) administered prior to discharge followed by a second injection one month later. The central hypothesis is that hospital-administered, long-acting injectable naltrexone, when compared to daily oral naltrexone, will reduce alcohol use in the days immediately following hospitalization. This reduced consumption, we hypothesize, will be followed by improved engagement in substance abuse treatment.

Primary Aim: Demonstrate the feasibility of the proposed recruitment methods and study design. This aim comprises two measures with corresponding goals: (1) Recruitment/enrollment-with a recruitment goal of 50 eligible and consenting subjects in an 8 month time period, and (2) Follow-up data collection with a goal of post-hospitalization follow-up data on no less than 70% of enrolled subjects.

Secondary Aims: As a pilot feasibility study, we may not anticipate sufficient power to attain statistical significance on patient-oriented outcome measures. However, it will be important for us to consider and to evaluate pertinent outcomes and potential moderators in order to (1) develop and fine-tune study design, and (2) determine effect sizes for primary outcomes so that we may calculate appropriate sample sizes for future larger study. As such, the secondary aims for the current study are:

1. To compare injectable naltrexone study to oral naltrexone in terms of attendance to recommended outpatient substance abuse treatment. We hypothesize that injectable naltrexone will be associated with improved likelihood of attending initial visits for substance abuse treatment.
2. To compare study arms in terms of ongoing alcohol consumption. We hypothesize that (1) improved medication adherence in the oral naltrexone arm and (2) assignment to injectable naltrexone will be associated with reduced alcohol consumption (number of heavy drinking days in the past 14 days) following hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* diagnostic criteria for alcohol dependence or abuse
* women of childbearing potential who have a negative screening urine pregnancy test and are willing to use reliable birth control methods throughout the duration of the study

Exclusion Criteria:

* active or recently active (less than 1 year) opioid dependence or daily use of opioid analgesics
* acute hepatitis or liver failure
* pregnancy
* women who are currently breastfeeding
* active suicidality
* inability to provide written informed consent as determined by study comprehension questions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall T Brown, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin - Department of Family Medicine, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 9 participants who didn't receive medication were discharged from the hospital before they could get medication.
  Therefore, only 45 , out of 54 participants got the medication.
Period: Overall Study
Arm/Group | Oral Naltrexone | Injectable Naltrexone
Started | 23 | 22 (1 received oral in error thus randomized.)
Lost to 14 Day Follow up | 6 | 2
Lost to 45 Day Follow up | 1 | 1
Completed | 16 | 19
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Population: Out of 54 enrolled participants, 9 participants were discharged before they could get medication.
  23 participants received oral naltrexone, 22 participants received injectable naltrexone (1 received oral in error and was analyzed as randomized).
  Total 45 participants received intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Naltrexone | Injectable Naltrexone | Total
Number analyzed (Participants) | 23 | 22 | 45
Age, Categorical [Count of Participants; unit: Participants] — Population: Oral naltrexone: 4 did not receive intervention Injectable natrexone: 5 did not receive intervention
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 15 | 16 | 31
    >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Oral naltrexone: 4 did not receive intervention Injectable natrexone: 5 did not receive intervention
  years | 50.9 (14.5) | 48.3 (12.9) | 49.5 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Oral naltrexone: 4 participants did not receive intervention Injectable naltrexone: 5 did not receive intervention
  Participants
    Female | 1 | 21 | 22
    Male | 22 | 1 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Oral naltrexone: 4 did not receive intervention Injectable natrexone: 5 did not receive intervention. Not receiving intervention medication was related to discharge from the hospital prior to receiving.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 3 | 2 | 5
    White | 20 | 20 | 40
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 | 45

OUTCOME MEASURES:

1. Primary Outcome: Retention Rate: Percentage of Participants Attended an Initial Behavioral Treatment Visit Within 2 Weeks of Hospital Discharge.
Description: Retention rate was measured in terms of percentage of participants attended an initial behavioral treatment visit within 2 weeks of hospital discharge.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Oral Naltrexone: enrolled and received oral naltrexone
- Injectable Naltrexone: enrolled and received injectable naltrexone
Arm/Group | Oral Naltrexone | Injectable Naltrexone
Number analyzed (Participants) | 23 | 22
Participants | 23 | 22
Statistical Analysis 1: Comparison: Oral Naltrexone vs Injectable Naltrexone; Test type: Superiority; Odds Ratio (OR) = 1.71, 95% CI 2-sided [0.35 to 9.98]

2. Secondary Outcome: Percentage of Patients Attended Recommended Outpatient Substance Abuse Treatment
Description: Attendance to recommended outpatient substance abuse treatment will be compared between injectable naltrexone group and oral naltrexone group. Keeping patients engaged in treatment is desirable and is known to improve addiction-related outcomes.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Oral Naltrexone: an initial 50 mg oral dose of naltrexone prior to hospital discharge plus a 30-day prescription for oral naltrexone
  Naltrexone: Naltexone was chosen for this study because naltrexone is the only medication available in both oral daily and injectable monthly formulations, which will allow the study to examine issues around medication adherence.
  Among those who were randomized (n=54), 64.8% (n=35) received a study medication and completed all follow-ups. Among those received a study medication and were proactively followed (n=45), 77% completed all follow-ups.
- Injectable Naltrexone: a single 380 mg intramuscular injection of naltrexone (duration of action = 30 days)prior to hospital discharge followed by a second injection one month later.
  Naltrexone: Naltexone was chosen for this study because naltrexone is the only medication available in both oral daily and injectable monthly formulations, which will allow the study to examine issues around medication adherence.
  Among those who were randomized (n=54), 64.8% (n=35) received a study medication and completed all follow-ups. Among those received a study medication and were proactively followed (n=45), 77% completed all follow-ups.
Arm/Group | Oral Naltrexone | Injectable Naltrexone
Number analyzed (Participants) | 23 | 22
Participants | 19 | 18

3. Secondary Outcome: Percentage of Participants Adhered to Medication
Description: Medication adherence was measured as percentage of participants who took ≥ 80% of daily naltrexone doses determined via pill counts. Adherence of daily medication will predict treatment engagement following hospital discharge.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Oral Naltrexone: an initial 50 mg oral dose of naltrexone prior to hospital discharge plus a 30-day prescription for oral naltrexone
  Naltrexone: Naltexone was chosen for this study because naltrexone is the only medication available in both oral daily and injectable monthly formulations, which will allow the study to examine issues around medication adherence.
  Among those who were randomized (n=54), 64.8% (n=35) received a study medication and completed all follow-ups. Among those received a study medication and were proactively followed (n=45), 77% completed all follow-ups. 62% of injection group and 61% of oral group met study definition of adherence
- Injectable Naltrexone: a single 380 mg intramuscular injection of naltrexone (duration of action = 30 days)prior to hospital discharge followed by a second injection one month later.
  Naltrexone: Naltexone was chosen for this study because naltrexone is the only medication available in both oral daily and injectable monthly formulations, which will allow the study to examine issues around medication adherence.
  Among those who were randomized (n=54), 64.8% (n=35) received a study medication and completed all follow-ups. Among those received a study medication and were proactively followed (n=45), 77% completed all follow-ups. 62% of injection group and 61% of oral group met study definition of adherence
Arm/Group | Oral Naltrexone | Injectable Naltrexone
Number analyzed (Participants) | 23 | 22
Participants | 14 | 14

4. Secondary Outcome: Ongoing Alcohol Consumption
Description: To compare study arms in terms of ongoing alcohol consumption. We hypothesize that (1) improved medication adherence in the oral naltrexone arm and (2) assignment to injectable naltrexone will be associated with reduced alcohol consumption (number of heavy drinking days in the past 14 days) following hospital discharge.
Time Frame: 12 months
Measure: Mean (Inter-Quartile Range); unit: Total drinks
Arm/Group | Oral Naltrexone | Injectable Naltrexone
Number analyzed (Participants) | 23 | 22
Total drinks | 136.5 [1 to 364] | 114.5 [0 to 308]

ADVERSE EVENTS:
Time Frame: from September 5, 2013 to April 20, 2015, for a total accrual time of 19 months
Arm/Group | Oral Naltrexone | Injectable Naltrexone
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 1/23 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Naltrexone (N=23) | Injectable Naltrexone (N=22)
depression (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes